CLINICAL TRIAL: NCT02066532
Title: Phase I/II Trial of Ruxolitinib in Combination With Trastuzumab in Metastatic HER2 Positive Breast Cancer
Brief Title: Ruxolitinib in Combination With Trastuzumab in Metastatic HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dawn L. Hershman (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Dawn L. Hershman, Professor of Medicine and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAM1906; 5U01CA168426 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-02-19 (Estimated); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Breast Cancer; Breast Carcinoma; HER-2 Positive Breast Cancer
Keywords: Breast Neoplasms; Breast Cancer; Breast Carcinoma; Breast tumors; Cancer of the Breast; Malignant tumor of the breast; HER2 positive; erythroblastosis virus oncogene B-2 (erbB-2); Metastatic Breast Cancer; Secondary Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ruxolitinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib/Trastuzumab (Experimental): Jakafi (Ruxolitinib) and Trastuzumab (Herceptin) - 21 day cycle until disease progression
  Interventions: Drug: Ruxolitinib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Ruxolitinib — 25 mg bid, 20 mg bid, 15 mg bid, or 10 mg bid, (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Jakafi
Drug: Trastuzumab — 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Ruxolitinib in combination with Trastuzumab in treatment of HER2 positive metastatic breast cancer. Ruxolitinib (Jakafi) is an Food and Drug Administration (FDA) approved treatment for myelofibrosis (a disease of the bone marrow), but its safety and efficacy in breast cancer patients is not known. Trastuzumab (Herceptin) is an FDA-approved treatment for HER2 positive breast cancer. The safety and efficacy of both treatments given in combination is not known. It is hypothesized that Ruxolitinib in combination with Trastuzumab will demonstrate efficacy in treating Metastatic HER2 Positive Breast Cancer subjects, and will have a tolerable safety profile in this patient population.

DETAILED DESCRIPTION:
Breast cancer is the most common female cancer and the second most common cause of cancer death in women. Approximately 1,150,000 cases and 410,000 deaths from breast cancer occur annually worldwide, and, in the U.S., there are an estimated 184,450 new cases and 40,480 deaths from breast cancer every year. The vast majority of patients who die from breast cancer succumb to metastatic disease. The human epidermal growth factor receptor type 2 gene (HER2) is amplified in 20% to 30% of breast cancers.

HER2+ breast cancers are associated with earlier recurrence and shorter overall survival and are associated with other adverse prognostic markers, such as high tumor grade, high rates of cell proliferation, increased nodal metastases, and relative resistance to certain types of chemotherapy. The HER family of receptors is a group of related transmembrane receptor tyrosine kinases that regulate normal cell survival, proliferation, differentiation, and migration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease. Locally recurrent disease must not be amenable to any local treatment with curative intent. Metastatic disease must be demonstrated either radiographically or histologically.
* Primary tumors and/or metastatic lesions must demonstrate HER2-neu overexpression, per the 2013 recommendations, i.e. immunohistochemistry (IHC 3+) or amplification by in situ hybridization based on the following:

  1. Single-probe average HER2 copy number ≥6.0 signals/cell
  2. Dual-probe HER2/Chromosome 17 centromere (CEP17) ratio ≥2.0 with an average HER2 copy number ≥4.0 signals/cell
  3. Dual-probe HER2/CEP17 ratio ≥2.0 with an average HER2 copy number <4.0 signals/cell
  4. Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number > 6.0 signals/cell
* Patients should have progressed on at least two lines of HER2-directed therapy in the metastatic setting, and prior therapy for metastatic disease should include both pertuzumab and ado-trastuzumab unless contraindicated or declined by the patient.
* There is no upper limit on the number prior therapies
* Patients may have measurable disease only, non-measurable disease only, or both (RECIST 1.1). Concomitant treatment with bone-targeted therapies such as Receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitors or bisphosphonates is allowed. It is anticipated that most patients will have measurable disease, given the behavior of HER2+ metastatic breast cancer.
* Because no dosing or adverse event data are currently available on the use of ruxolitinib in combination with trastuzumab in patients <18 years of age, children are excluded from this study.
* Women and men of all races and ethnic groups are eligible for this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky equal to or greater than 60)
* Left ventricular ejection fraction greater than or equal to 50 percent by transthoracic echocardiography or multi-gated acquisition scan (MUGA) within 28 days prior to the first dose of the study drug.
* The subject has a baseline corrected QT interval less than or equal to 480ms.
* Patients must have normal organ and marrow function as defined below:

  1. leukocytes greater than or equal to 3,000/microliter (mcL).
  2. absolute neutrophil count greater than or equal to 1,500/mcL.
  3. platelets greater than or equal to 100,000/mcL.
  4. hemoglobin greater than or equal to 9 g/dL.
  5. total bilirubin less than or equal to 1.5 times the upper limit of normal.
  6. Aspartate Aminotransferase (AST/SGOT)/ Alanine Aminotransferase (ALT/SGPT) less than or equal to 2.5 time institutional upper limit of normal.
  7. Serum creatinine less than or equal to 1.5 times the upper limit of normal or calculated creatinine clearance greater than or equal to 60 mL/min.
* Women of childbearing potential and men must use adequate contraception prior to study entry and for the duration of study participation. Contraception should continue to be used for a minimum of 5 mean half-lives after the last dose of study drugs (mean Trastuzumab half-life at 6 mg/kg 16 days; mean half-life Ruxolitinib: 3 hours)
* Patient is able to swallow, retain, and absorb oral medication.
* Informed Consent. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy, hormonal therapy, or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Patients who are receiving any other investigational agents or have received other investigational agents within 2 weeks or 5 half-lives of the compound or active metabolites, whichever is longer before the first dose of the study treatment.
* Patients who have previously been treated with an interleukin-6 (IL-6), Janus kinase (JAK) or Signal Transducers and Activators of Transcription (STAT) inhibitor for any indication, such as ruxolitinib or tocilizumab.
* The subject has untreated, symptomatic, or progressive brain metastases. History of Central Nervous System (CNS) metastases or cord compression is allowable if patient has been clinically stable for at least 6 weeks since completion of definitive treatment and is off steroids without symptoms for at least 28 days.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or trastuzumab.
* The effects of ruxolitinib on the developing human fetus are unknown. For this reason and because Janus kinase 2 (JAK2) inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the principal investigator immediately.
* Patients receiving any medications or substances that are strong inhibitors of cytochrome P450 (CYP450) 3A4 isoenzyme are ineligible. Patients must be off the strong inhibitor for at least 1 week prior to being deemed eligible.
* Patients may not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements.
* Patients must not have clinically significant cardiovascular disease (New York Heart Association Class III or IV heart failure), uncontrolled clinically significant atrial or ventricular cardiac arrhythmias, or any of the following within the past 6 months: myocardial infarction, new evidence of transmural infarction on electrocardiogram (ECG), unstable angina, coronary angioplasty.
* Pregnant women are excluded from this study because ruxolitinib is a Class C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding must be discontinued if the mother is treated with ruxolitinib. These potential risks also apply to trastuzumab, which can cause fetal harm when administered to a pregnant woman.
* Active Infections. Patients with known active infections with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis B (HBV), and hepatitis C virus (HCV) infections will not be considered for this trial. HIV+ patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ruxolitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Testing for HIV or hepatitis is not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, MS, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Hospital-Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — http://hiccc.columbia.edu/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 32 participants enrolled. The first 10 enrolled participated in phase I. Nine of the ten participants enrolled during phase I continued to phase II. An additional 22 participants enrolled in phase II. Five did not meet eligibility criteria, resulting in 26 allocated to intervention.
Groups:
- Ruxolitinib (25mg)/Trastuzumab: Ruxolitinib: 25 mg bid (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
- Ruxolitinib (20mg)/ Trastuzumab: Ruxolitinib: 20 mg bid (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
- Ruxolitinib (15 mg)/ Trastuzumab: Ruxolitinib: 15 mg bid (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
- Ruxolitinib (10 mg)/ Trastuzumab: Ruxolitinib:10 mg bid, (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
Period: Phase I
Arm/Group | Ruxolitinib (25mg)/Trastuzumab | Ruxolitinib (20mg)/ Trastuzumab | Ruxolitinib (15 mg)/ Trastuzumab | Ruxolitinib (10 mg)/ Trastuzumab
Started | 9 | 1 | 0 | 0
Completed | 9 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Ruxolitinib (25mg)/Trastuzumab | Ruxolitinib (20mg)/ Trastuzumab | Ruxolitinib (15 mg)/ Trastuzumab | Ruxolitinib (10 mg)/ Trastuzumab
Started | 27 | 0 | 0 | 0
Completed | 26 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As only one participant was included in the Phase 1: Ruxolitinib (20mg)/ Trastuzumab arm, they are not represented in the baseline analysis population in an effort to protect their confidentiality.
Groups:
- Phase 1 and Phase 2: Ruxolitinib/Trastuzumab (25 mg): Ruxolitinib: 25 mg bid (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
Arm/Group | Phase 1 and Phase 2: Ruxolitinib/Trastuzumab (25 mg)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: Years] | 56 [32 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Indian | 2
  Black | 6
  White | 15
  Unknown/other | 3
Region of Enrollment [Number; unit: participants]
  United States | 26
Hormone receptor positive [Count of Participants; unit: Participants] | 19
Hormone receptor negative [Count of Participants; unit: Participants] | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scale describes a participant's level of function regarding their ability to care for themselves, daily activity, and physical ability. Grades (scores) range from 0 (Fully active) to 5 (death).
  Participants
    ECOG Score 0 | 14
    ECOG Score 1 | 12
Metastatic at time of diagnosis [Count of Participants; unit: Participants] | 14
Post-menopausal [Count of Participants; unit: Participants] | 24
Prior systemic therapy [Median (Full Range); unit: number of prior regimens] | 4.5 [1 to 10]
Prior pertuzumab [Count of Participants; unit: Participants] | 23
Prior ado-trastuzumab emtansine [Count of Participants; unit: Participants] | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ruxolitinib in Combination With Trastuzumab (Phase I)
Description: The maximum tolerated dose (MTD) combination is defined as the dose combination associated with a target probability of dose limiting toxicity (DLT) of 0.25. A dose-limiting toxicity is defined as the MTD with DLTs defined as any grade 3 non-hematologic toxicities despite maximal supportive care or any grade 4 hematologic toxicity. The MTD will be estimated using the time to event continual reassessment method (TITE-CRM). The TITE-CRM will use an empirical dose-toxicity model, with a sample size of 10. The dose-toxicity model is calibrated such that the method will eventually select a dose that yields between 16% and 34% DLT.
Time Frame: Up to 15 weeks
Measure: Number; unit: milligrams
Arm/Group | Ruxolitinib/Trastuzumab
Number analyzed (Participants) | 10
milligrams | 25

2. Primary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Progression free survival (PFS) will be measured every 3 cycles (9 weeks of treatment +/- 4 days). PFS will be defined as the time from patient registration until objective or disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 24 weeks
Population: Phase II participants
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Ruxolitinib/Trastuzumab: Ruxolitinib: 25 mg bid (oral, twice a day) on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
Arm/Group | Ruxolitinib/Trastuzumab
Number analyzed (Participants) | 26
Weeks | 8.3 [7.1 to 13.9]

3. Secondary Outcome: Objective Response Rate (Phase II)
Description: Participants will be reviewed at 24 weeks to determine the objective response rate, which is defined as the number of participants with a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Time Frame: Up to 24 weeks
Population: Phase II participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib/Trastuzumab
Number analyzed (Participants) | 26
Participants | 1

4. Secondary Outcome: Number of Participants With Adverse Events (Phase II)
Description: All phase II participants were evaluated for toxicity from the time of their first treatment with the study drugs. The frequency of subjects experiencing toxicities will be tabulated using the Canter Therapies Evaluation Program (CTEP) Active Version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 4.0).
Time Frame: Up to 6 years
Population: Phase II participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib/Trastuzumab
Number analyzed (Participants) | 26
Participants | 26

5. Secondary Outcome: Clinical Benefit Ratio (CBR) (Phase II)
Description: CBR defined as complete response, partial response, or stable disease for >24 weeks in the phase II portion
Time Frame: 24 weeks
Population: Phase II participants
Measure: Number; unit: participants
Arm/Group | Ruxolitinib/Trastuzumab
Number analyzed (Participants) | 26
participants | 4

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: As only one participant was included in the Phase 1: Ruxolitinib (20mg)/ Trastuzumab arm, they are not represented in the adverse event tables in an effort to protect their confidentiality.
Groups:
- Phase 1 and 2: Ruxolitinib/Trastuzumab (25 mg): Ruxolitinib: 25 mg bid on days 1 through 21 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Trastuzumab: 6 mg/kg every 3 weeks (cycle = 21 days). If no trastuzumab > 28 days, patients will be initially re-loaded at 8 mg/kg, then 6 mg/kg.
Arm/Group | Phase 1 and 2: Ruxolitinib/Trastuzumab (25 mg)
All-Cause Mortality (participants affected / at risk) | 4/26
Serious Adverse Events (participants affected / at risk) | 8/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 and 2: Ruxolitinib/Trastuzumab (25 mg) (N=26)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Wound Infection (Infections and infestations) | 1
Nervous System Disorder (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chest Pain (Cardiac disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3
Thromboembolic Event (Vascular disorders) | 1
Seizure (Nervous system disorders) | 1
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Musculoskeletal and connective tissue disorders) | 2
Upper respiratory infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 and 2: Ruxolitinib/Trastuzumab (25 mg) (N=26)
Pain in extremity (General disorders) | 1
Muscle weakness, upper limb (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Eye Disorder (Eye disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increase (Blood and lymphatic system disorders) | 5
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 4
Allergic rhinitis (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ascites (General disorders) | 1
Aspartate aminotransferase increase (Blood and lymphatic system disorders) | 8
Bloating (Gastrointestinal disorders) | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5
Blood bilirubin increased (Blood and lymphatic system disorders) | 1
Blurred vision (Eye disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
CD4 lymphocytes decrease (Blood and lymphatic system disorders) | 1
Chest pain- cardiac (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Cholesterol high (Blood and lymphatic system disorders) | 2
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (General disorders) | 2
Creatinine increase (Blood and lymphatic system disorders) | 4
Cystitis noninfective (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (General disorders) | 5
Dry eye (Eye disorders) | 1
Dry mouth (General disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
Ejection fraction decreased (Cardiac disorders) | 1
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1
Epistaxis (General disorders) | 1
Fall (General disorders) | 1
Fatigue (General disorders) | 10
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (Nervous system disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders, other (Gastrointestinal disorders) | 2
Gastroparesis (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (General disorders) | 3
Heart failure (Cardiac disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Hoarseness (General disorders) | 1
Hot flashes (General disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 3
Hyperkalemia (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 4
Hypocalcemia (Blood and lymphatic system disorders) | 3
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 2
Hypoxia (General disorders) | 2
Infections and infestations, other (Infections and infestations) | 2
Infusion related reaction (General disorders) | 1
Insomnia (Nervous system disorders) | 1
Localized edema (General disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 10
Non-cardiac chest pain (General disorders) | 2
Oral pain (General disorders) | 1
Pain (General disorders) | 2
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Premature menopause (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rectal mucositis (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 2
Sore throat (Gastrointestinal disorders) | 1
Spasticity (Musculoskeletal and connective tissue disorders) | 1
Toothache (General disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Tumor pain (General disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (General disorders) | 4
Weight loss (General disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 9
General disorders and administration site conditions - Other, specify (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02066532/Prot_SAP_000.pdf